CLINICAL TRIAL: NCT00005549
Title: Isocyanate Antigens and T Cells That Cause Asthma
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 5093; R01HL062622 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To investigate whether isocyanate-induced asthma is dependent on isocyanate antigen-driven T-cell mediated, airway inflammation.

DETAILED DESCRIPTION:
BACKGROUND:

Isocyanates are a group of highly reactive widely used low-molecular weight chemicals, and are the most commonly reported cause of occupation asthma in developed countries. Yet, the mechanisms by which isocyanates cause asthma are not well defined.

DESIGN NARRATIVE:

The study investigates isocyanate antigen-driven T-cell responses in vitro-, following in vivo exposure using patient samples acquired through collaboration with ongoing field epidemiological and clinical studies. The study compares isocyanate antigen-reactive T-cells from primary exposure sites (skin/lung) with those from blood, to evaluate potential routes of sensitization and identify diagnostic indicators of isocyanate sensitivity/susceptibility. Specifically, the study : generates and characterizes hexamethylene diisocyanate (HDI) antigens including isocyanate metabolites, and isocyanate conjugated t normal human and foreign proteins; evaluates the T-cell antigenicity of the HDI antigens, based on blood and lung lymphocyte proliferation, cytokine production, and phenotype in order to identify the molecular form of HDI that initiates airway cytokine production in asthma patients; establishes T-cell lines from the skin, lung and peripheral blood of HDI asthma patients and characterizes the phenotype, antigen specificity, cytokine production and TCR expression of isocyanate responsive T-cells in these different compartments; compares isocyanate responsive of T-cells found in the skin, lung and blood and correlates with clinical sensitivity to determine characteristics associated with exposure and sensitization leading to clinical asthma.

The study was renewed in FY 2002 to extend follow-up and analysis through March 2007.

ELIGIBILITY:
No eligibility criteria

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-01; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Wisnewski — Yale University

REFERENCES:
- [Background] Wisnewski AV, Srivastava R, Herick C, Xu L, Lemus R, Cain H, Magoski NM, Karol MH, Bottomly K, Redlich CA. Identification of human lung and skin proteins conjugated with hexamethylene diisocyanate in vitro and in vivo. Am J Respir Crit Care Med. 2000 Dec;162(6):2330-6. doi: 10.1164/ajrccm.162.6.2002086. PMID 11112159
- [Background] Wisnewski AV, Cain H, Magoski N, Wang H, Holm CT, Redlich CA. Human gamma/delta T-cell lines derived from airway biopsies. Am J Respir Cell Mol Biol. 2001 Mar;24(3):332-8. doi: 10.1165/ajrcmb.24.3.4325. PMID 11245633
- [Background] Redlich CA, Stowe MH, Coren BA, Wisnewski AV, Holm CT, Cullen MR. Diisocyanate-exposed auto body shop workers: a one-year follow-up. Am J Ind Med. 2002 Dec;42(6):511-8. doi: 10.1002/ajim.10143. PMID 12439874
- [Background] Wisnewski AV, Liu Q, Miller JJ, Magoski N, Redlich CA. Effects of hexamethylene diisocyanate exposure on human airway epithelial cells: in vitro cellular and molecular studies. Environ Health Perspect. 2002 Sep;110(9):901-7. doi: 10.1289/ehp.02110901. PMID 12204825
- [Background] Liu Q, Wisnewski AV. Recent developments in diisocyanate asthma. Ann Allergy Asthma Immunol. 2003 May;90(5 Suppl 2):35-41. doi: 10.1016/s1081-1206(10)61647-x. PMID 12772950
- [Background] Wisnewski AV, Stowe MH, Cartier A, Liu Q, Liu J, Chen L, Redlich CA. Isocyanate vapor-induced antigenicity of human albumin. J Allergy Clin Immunol. 2004 Jun;113(6):1178-84. doi: 10.1016/j.jaci.2004.03.009. PMID 15208602
- [Background] Wisnewski AV, Herrick CA, Liu Q, Chen L, Bottomly K, Redlich CA. Human gamma/delta T-cell proliferation and IFN-gamma production induced by hexamethylene diisocyanate. J Allergy Clin Immunol. 2003 Sep;112(3):538-46. doi: 10.1016/s0091-6749(03)01865-7. PMID 13679813
- [Background] Wisnewski AV, Liu Q, Liu J, Redlich CA. Glutathione protects human airway proteins and epithelial cells from isocyanates. Clin Exp Allergy. 2005 Mar;35(3):352-7. doi: 10.1111/j.1365-2222.2005.02185.x. PMID 15784115